CLINICAL TRIAL: NCT06719674
Title: Impact of Diode Laser as an Adjunct to Professional Mechanical Plaque Removal (PMPR) in Patients With Periodontitis: A Randomized Clinical Trial
Brief Title: Diode Laser as an Adjunct to Professional Mechanical Plaque Removal
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Sulaimani (Other)
Collaborators: University of Dundee (Other); Sulaimany Polytechnic university (Other)
Responsible Party: Principal Investigator, Sarhang Gul, Asst. Prof. Dr., University of Sulaimani
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USulaimani/SGUL
Record Dates: First submitted 2024-12-01; First posted 2024-12-06 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis; Pocket, Periodontal
Keywords: Non surgical periodontal therapy; Diode laser; Salivary biomarkers
MeSH Terms: conditions — Periodontitis; Periodontal Pocket | interventions — Lasers; Photochemotherapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Professional Mechanical Plaque Removal + Laser (Experimental): The patients will be treated in accordance with treatment guidelines for Stage III periodontitis issued by the European Federation of Periodontology. At baseline, oral hygiene instructions were given together with supra- and subgingival professional mechanical plaque removal (PMPR) using a combination of the ultrasonic scaler and hand instruments plus diode laser, according to the clinical situation. After completing treatment, patients will be asked to return at 1 month for review and again at 3 months to repeat the measurement of clinical parameters and collection of the saliva samples.
  Interventions: Procedure: Professional mechanical plaque removal and Laser
- Professional Mechanical Plaque Removal (Active Comparator): The patients will be treated in accordance with treatment guidelines for Stage III periodontitis issued by the European Federation of Periodontology (13). At baseline, oral hygiene instructions were given together with supra- and subgingival professional mechanical plaque removal (PMPR) using a combination of the ultrasonic scaler and hand instruments, according to the clinical situation. After completing treatment, patients will be asked to return at 1 month for review and again at 3 months to repeat the measurement of clinical parameters and collection of the saliva samples.
  Interventions: Procedure: Professional mechanical plaque removal

INTERVENTIONS:
Procedure: Professional mechanical plaque removal and Laser — A diode laser will be used as an adjunct to mechanical plaque removal.
  Other Names: EPIC 10S Soft Tissue Diode Laser; Photodynamic therapy
  Arms: Professional Mechanical Plaque Removal + Laser
Procedure: Professional mechanical plaque removal — The patients will be treated in accordance with treatment guidelines for Stage III periodontitis issued by the European Federation of Periodontology (13). At baseline, oral hygiene instructions were given together with supra- and subgingival professional mechanical plaque removal (PMPR) using a combination of the ultrasonic scaler and hand instruments, according to the clinical situation. After completing treatment, patients will be asked to return at 1 month for review and again at 3 months to repeat the measurement of clinical parameters and collection of the saliva samples.
  Arms: Professional Mechanical Plaque Removal

SUMMARY:
This study will utilize diode laser to determine its effects on improving periodontal parameters and inflammatory biomarkers, comparing with conventional treatment alone, and evaluate its effectiveness in improving periodontal disease's clinical parameters. Several studies have compared the effects of lasers and conventional periodontal treatment, comparing only its microbiological and clinical parameter levels and therapy to determine their effectiveness in key periodontal pathogens eradication and their effects on improving the clinical parameters of periodontal disease, in this study, salivary biomarkers will be collected and assessed to do a comparison between two treatment modalities. To the best of our knowledge, this is the first study to examine the effect of diode lasers on salivary biomarker levels.

DETAILED DESCRIPTION:
Periodontitis is an inflammatory disease caused by dental biofilm that provokes a chronic immune-inflammatory response that eventually causes the gradual loss of the periodontal tissues supporting the teeth. The evaluation of the disease is determined by clinical attachment loss (CAL), probing pocket depth (PPD), bleeding on probing (BOP), and the assessment of alveolar bone radiographically. Periodontal disease is a well-established disease that certainly impacts the general well-being of patients. It is closely linked to poor oral health-related quality of life, particularly in patients with moderate to severe periodontitis.

Moreover, a comprehensive study has demonstrated a direct correlation between the severity of the disease, as indicated by higher staging and grading, and an increased likelihood of tooth loss. The primary goal of periodontal therapy is to prevent or arrest the spread of the periodontal infection. The standard treatment approaches involve non-surgical or surgical periodontal therapy. Mechanical instrumentation (professional mechanical plaque removal - PMPR) is the gold standard in treating periodontal diseases; however, it can be challenging to reach and effectively remove calculus and bacterial deposits in the irregular and furcation areas. Therefore, an adjunctive aid like systemic or local antibiotics is sometimes necessary to be administered. Nevertheless, they have many adverse effects and it is also important to reduce the use of systemic antibiotics given the increases in antimicrobial resistance that occur globally.

Another adjunctive aid such as laser has been introduced to the field of periodontology to achieve bacterial eradication with minimum side effects. The term "laser" is derived from the abbreviation "light amplification by stimulated emission of radiation." A laser is a device that produces a well-aligned light beam that is well concentrated, which can maintain its narrowness across a significant distance and be firmly focused. When targeted towards tissues, many interactions occur. The behavior of laser light, including absorption, reflection, transmission, and scattering, is influenced by the laser's wavelength and the tissue's properties.

The primary objective of adjunctive laser use in periodontal therapy is to eliminate the inflamed and necrotic tissues located within the periodontal sulcus. The use of lasers is a contemporary adjunctive to traditional periodontal therapy for treating periodontitis. The alleged benefits of laser therapy include enhanced accessibility to root surfaces, more reliable control of bleeding, and better patient acceptability as it eliminates the requirement for conventional surgical flaps and sutures.

ELIGIBILITY:
Inclusion Criteria:

* Patient with periodontitis.
* Patients having at least 3 teeth with PPD of 5 mm and above.

Exclusion Criteria:

* Patients with diabetes
* Patients on medication with an inhibitory or promoting effect on periodontal healing, including anticoagulants, anti-inflammatory drugs.
* Patients received antibiotics within the last three months.
* Pregnant or nursing women
* Patients receiving periodontal therapy within the last 3 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction in probing pocket depth (mm) | 3 months
  Probing pocket depth determined from the gingival margin to the base of the pocket at six sites per tooth.

SECONDARY OUTCOMES:
Biomarkers level in pg/ML: (interleukin (IL)-1beta), Matrix metalloproteinases (MMP 8) and (TIMP), RANK. | 3 months
  The analysis of salivary biomarkers involves different techniques depending on the biomarker of interest, including Enzyme-Linked Immunosorbent Assay (ELISA): A widely used method for detecting proteins, hormones, and cytokines in saliva.

CONTACTS AND LOCATIONS:
Overall Officials: Sarhang S Gul, Principal Investigator — University of Sulaimani
Locations (1):
- College of Dentistry, University of Sulaimani, Sulaymaniyah, Iraq

IPD SHARING:
Plan to Share IPD: No
The data will be available upon reasonable request by the principal investigator.

REFERENCES:
- [Background] Papapanou PN, Sanz M, Buduneli N, Dietrich T, Feres M, Fine DH, Flemmig TF, Garcia R, Giannobile WV, Graziani F, Greenwell H, Herrera D, Kao RT, Kebschull M, Kinane DF, Kirkwood KL, Kocher T, Kornman KS, Kumar PS, Loos BG, Machtei E, Meng H, Mombelli A, Needleman I, Offenbacher S, Seymour GJ, Teles R, Tonetti MS. Periodontitis: Consensus report of workgroup 2 of the 2017 World Workshop on the Classification of Periodontal and Peri-Implant Diseases and Conditions. J Periodontol. 2018 Jun;89 Suppl 1:S173-S182. doi: 10.1002/JPER.17-0721. PMID 29926951
- [Background] Shaddox LM, Walker CB. Treating chronic periodontitis: current status, challenges, and future directions. Clin Cosmet Investig Dent. 2010 Aug 11;2:79-91. Print 2010. PMID 23662085
- [Background] Ravida A, Qazi M, Rodriguez MV, Galli M, Saleh MHA, Troiano G, Wang HL. The influence of the interaction between staging, grading and extent on tooth loss due to periodontitis. J Clin Periodontol. 2021 May;48(5):648-658. doi: 10.1111/jcpe.13430. Epub 2021 Mar 19. PMID 33484162
- [Background] Ciantar M. Time to shift: from scaling and root planing to root surface debridement. Prim Dent J. 2014 Aug;3(3):38-42. doi: 10.1308/205016814812736592. PMID 25198637
- [Background] Keeney KM, Yurist-Doutsch S, Arrieta MC, Finlay BB. Effects of antibiotics on human microbiota and subsequent disease. Annu Rev Microbiol. 2014;68:217-35. doi: 10.1146/annurev-micro-091313-103456. Epub 2014 Jun 2. PMID 24995874
- [Background] Nevins ML, Camelo M, Schupbach P, Kim SW, Kim DM, Nevins M. Human clinical and histologic evaluation of laser-assisted new attachment procedure. Int J Periodontics Restorative Dent. 2012 Oct;32(5):497-507. PMID 22754897
- [Background] Luke AM, Mathew S, Altawash MM, Madan BM. Lasers: A Review With Their Applications in Oral Medicine. J Lasers Med Sci. 2019 Fall;10(4):324-329. doi: 10.15171/jlms.2019.52. Epub 2019 Oct 1. PMID 31875126
- [Background] Jha A, Gupta V, Adinarayan R. LANAP, Periodontics and Beyond: A Review. J Lasers Med Sci. 2018 Spring;9(2):76-81. doi: 10.15171/jlms.2018.16. Epub 2018 Mar 20. PMID 30026890
- [Background] Bechir ES. The Clinical and Microbiological Effects of LANAP Compared to Scaling and Root Planing Alone in the Management of Periodontal Conditions. Diagnostics (Basel). 2023 Jul 22;13(14):2450. doi: 10.3390/diagnostics13142450. PMID 37510194
- [Background] Cobb CM. Clinical significance of non-surgical periodontal therapy: an evidence-based perspective of scaling and root planing. J Clin Periodontol. 2002 May;29 Suppl 2:6-16. PMID 12010523
- [Background] Wassall RR, Preshaw PM. Clinical and technical considerations in the analysis of gingival crevicular fluid. Periodontol 2000. 2016 Feb;70(1):65-79. doi: 10.1111/prd.12109. PMID 26662483
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274